CLINICAL TRIAL: NCT05021939
Title: 2-dimensional Versus 3-dimensional Virtual Reality Game Training in Individuals With Benign Paroxysmal Positional Vertigo: A Randomized Controlled Study
Brief Title: 2-dimensional Versus 3-dimensional Virtual Reality Game Training in BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Aytül Özdil, Research Assistant, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2420-0107
Record Dates: First submitted 2021-08-17; First posted 2021-08-26 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Vertigo
Keywords: Benign paroxysmal positional vertigo; Dizziness; Virtual Reality; Vestibular Rehabilitation; Balance functions; Gait
MeSH Terms: conditions — Vertigo; Benign Paroxysmal Positional Vertigo; Dizziness

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant
Masking Description: The participants are blind to the treatment methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No treatment will be given to the control group. Evaluation will be done at the at the baseline and 8th week.
- 2-Dimensional Group (Experimental): In the 2-Dimensional Group, 2D VR gaming training in addition to traditional vestibular rehabilitation will be employed. In this group, the 'Verti-Go' game from the Playstation 4 VR gaming device will be played in 2D for 20-25 minutes, as well as vestibular therapy for 20-25 minutes. A total of 45-50 minutes will be given over the course of 8 weeks, 3 sessions per week. The intensity of treatment will rise with each session, depending on how well the patient cooperates. Evaluation will be done at the beginning and in the 8th week.
  Interventions: Other: 2-Dimensional Group
- 3-Dimensional Group (Experimental): In the 3-Dimensional Group, 3D VR gaming training in addition to traditional vestibular rehabilitation will be employed. In this group, the 'Verti-Go' game from the Playstation 4 VR gaming device with 3D glasses will be played for 20-25 minutes, as well as vestibular therapy for 20-25 minutes. A total of 45-50 minutes will be given over the course of 8 weeks, 3 sessions per week. The intensity of treatment will rise with each session, depending on how well the patient cooperates. Evaluation will be done at the beginning and in the 8th week.
  Interventions: Other: 3-Dimensional Group

INTERVENTIONS:
Other: 2-Dimensional Group — In the 2-Dimensional Group, 2D VR gaming training in addition to traditional vestibular rehabilitation will be employed. In this group, the 'Verti-Go' game from the Playstation 4 VR gaming device will be played in 2D for 20-25 minutes, as well as vestibular therapy for 20-25 minutes. A total of 45-50 minutes will be given over the course of 8 weeks, 3 sessions per week. The intensity of treatment will rise with each session, depending on how well the patient cooperates. Evaluation will be done at the beginning and in the 8th week.
  Arms: 2-Dimensional Group
Other: 3-Dimensional Group — In the 3-Dimensional Group, 3D VR gaming training in addition to traditional vestibular rehabilitation will be employed. In this group, the 'Verti-Go' game from the Playstation 4 VR gaming device with 3D glasses will be played for 20-25 minutes, as well as vestibular therapy for 20-25 minutes. A total of 45-50 minutes will be given over the course of 8 weeks, 3 sessions per week. The intensity of treatment will rise with each session, depending on how well the patient cooperates. Evaluation will be done at the beginning and in the 8th week.
  Arms: 3-Dimensional Group

SUMMARY:
Despite successful maneuver applications in the treatment of BPPV, complaints of balance problems and dizziness persist. Many studies supports the notion that virtual reality (VR) allowing visual-vestibular interaction with a large number of visual stimuli, contribute to successful outcomes in BPPV. VR applications using eye tracking algorithms and 'glasses' can be effective however. The research to date covers the VR technologies on the treatment of BPPV, however, there is no research comparing the effects of 2D and 3D VR gaming technologies with a control group. Therefore, this study aims to examine the effects of different virtual reality applications and vestibular rehabilitation on gait, reaction time, balance functions, activities of daily living, and quality of life in individuals with benign paroxysmal positional vertigo (BPPV) having residual dizziness and balance problems.

DETAILED DESCRIPTION:
The vestibular, visual, and somatosensory systems are all important in maintaining posture. Multiple structures of the central nervous system process and integrate afferents from these systems. The vestibular system is crucial for maintaining static and dynamic posture and balance. The vestibular system consists of two structures, peripheral and central. The peripheral vestibular system is located within the petrous bone and consists of the semicircular canals, utricle, and saccule in the inner ear that are sensitive to head movements. The semicircular canals consist of three parts: anterior, posterior and lateral semicircular canals. The semicircular canals, which are filled with a viscous fluid called endolymph, are located at right angles to each other and help to perceive the angular movements of the head. It transmits information about the peripheral vestibular system and head movements to the central systems via the vestibular nerve. In this way, it provides regulation of head, body, extremities and eye movements.

BPPV (Benign Paroxysmal Positional Vertigo) is a condition that affects the inner ear and is caused by semicircular canal dysfunction. Because the otoliths are placed in the semicircular canal and can impair their free movement, the anatomical placement of the canals is critical. BPPV is one of the most frequent peripheral vestibular illnesses with a prevalence of 20-40%. The first pathogenetic element is canalolithiasis, defined as the dissociation of the otoconia from the otolytic membrane and its free movement in the endolymph, which is seen in 80% of the patients. Cupulolithiasis is the occurrence of dizziness (vertigo) and nystagmus specific to the affected canal due to calcium carbonate crystals adhering to the canal. Because of its anatomical location, posterior semicircular canal BPPV is observed 80-90% of the time, lateral semicircular canal BPPV is seen 10-20% of the time, and anterior semicircular canal BPPV is less prevalent. BPPV often is treated with particle repositioning maneuvers once the involved canal is identified. These maneuvers are supposed to move otoconia particles out of the affected canal and back into the vestibule, where they dissolve.

Vestibular rehabilitation is another non-pharmacological intervention for BPPV. Vestibular rehabilitation can enhance general balance function, including gait, gaze, and postural stability, physical mobility, and function with activities of daily living, by integrating proprioceptive, visual, and residual vestibular function. Vestibular rehabilitation utilizes central neuroplasticity mechanisms to improve visuo-vestibular interactions and restore static and dynamic postural stability in situations where sensory input is conflicting. Vestibular rehabilitation includes adaptation, habituation, and substitution exercises. The adaptation exercises are based on the vestibular system's ability to change the magnitude of the vestibulo-ocular reflex (VOR) in response to a specific stimulus (head movement). Habituation exercises, in contrast to adaptation exercises, are based on the notion that frequent exposure to provoking stimuli such as head movements will reduce motion-provoked symptoms. Substitution exercises combine vision and somatosensory cues with vestibular cues to improve gaze and postural stability by enhancing central programming. Maneuvers are shown to be more successful than vestibular rehabilitation in the short term, although combining the two is useful for long-term functional recovery in BPPV. However, there is insufficient evidence to distinguish between different types of vestibular rehabilitation.

The positive impact of vestibular rehabilitation on balance is based on mechanisms related to the central nervous system's neural plasticity, and its goals are to promote visual stabilization, improve vestibular-visual interaction during head movements, thereby improving the standing and dynamic postural stability in conditions that produce conflicting sensory information, and decrease sensitivity to head movements. However, numerous aspects have been identified as having a detrimental impact on the outcome of vestibular rehabilitation, including poor exercise execution, the necessity for active efforts, and the patients' desire. Given the drawbacks associated with the time-consuming, repetitive, monotonous, and non-challenging aspects of vestibular rehabilitation, more efficient and cost-effective types of treatments were proposed as a potential alternative. Currently, virtual reality (VR) applications, can be outfitted with real-time simulations, interactive functions, and game features to allow for more motivated vestibular rehabilitation.

Many studies suggest that engaging virtual reality components can contribute to successful outcomes. It is claimed that it allows visual-vestibular interaction with a large number of visual stimuli, resulting in an optimal environment for better VR performance. It is suggested that this is due to the activation of target-oriented attention and the brain's neural network and that VR applications using eye-tracking algorithms and 'glasses' can be effective. In most of the studies, 2-dimensional systems (e.g. Nintendo Wii, Play station) has been used for the treatment of patients with BPPV. However, due to their proximity to the eye, head-mounted displays (3D VR gaming) may offer high-resolution images which make the users feel like they are a part of the computer-created environment. 3D technologies have been debated about their negative effects such as discomfort, visual fatigue, dizziness, headache, disorientation, motion sickness, which are indicative of VIMS (visually induced motion sickness). The most accepted explanation for VIMS is the classical conflict theory based on the mismatch between the visual, the proprioceptive, and the vestibular stimuli.

It is known that brief and sudden positional nystagmus associated with a change in head position relative to gravity may temporarily impair visual stability. The otolithic signal is created in response to the motion, which plays an important role in the perception of orientation and the direction of motion. Compensatory eye movement occurs after linear acceleration of the head, opposite in direction to the head movement, and is generated to stabilize the image of the target in coordination. The impact of dysfunction on the VOR in patients with chronic vestibular problems is associated with the inability to have a clear image of the target on the retina during head movements, resulting in blurred vision. According to these explanations, head movements while playing 3D VR gaming may pose a challenge (sensory mismatch) to the central nervous system, which then attempts to resolve the challenge. Habituation exercises included in the 3D VR gaming task might be beneficial in opposing over-reliance on a sensory modality, desensitizing patients to visual motion and visuo-vestibular conflict, and reducing associated symptoms.

It was proved out that accommodative facility has a tendency to increase after 2D and 3D VR gaming, but particular, the increasing tendency is greater after playing 3D VR gaming. It was explained that while playing a game, eyes are stimulated with stereoscopic images, and brightness change so that pupils remain under persistent stimulation. Therefore, the depth of a focus changes reversely and it results in visual training. In comparison to traditional 2D VR gaming technology, which does not provide depth to objects, 3D VR gaming technology may enable the perception of spatial depth. Additionally, it was proposed that the type of game (action vs. non-action) is important in 3D VR gaming. Especially, action game stimulates the overall parts of a brain, requiring multi-tasking skills and speed.

The research to date covers the VR technologies on the treatment of BPPV. However, to our knowledge, there is no research comparing the effects of 2D and 3D VR gaming technologies with a control group. Therefore, this study aims to examine the effects of different virtual reality applications and vestibular rehabilitation on gait, reaction time, balance functions, activities of daily living, and quality of life in individuals with benign paroxysmal positional vertigo (BPPV) having residual dizziness and balance problems.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of unilateral (either posterior or lateral semicircular canal) BPPV within the last 5 years,
2. Dix hallpike test negative (inactive BPPV),
3. Recurrent and persistent dizziness,
4. Balance problems,
5. Age 25-65 years old individuals will be included in the study.

Exclusion Criteria:

1. Episodic and secondary BPPV,
2. Anterior semicircular canal BPPV or multi-canal BPPV,
3. Coexisting vestibular disorders, including Meniere disease, vestibular neuritis, labyrinthitis and peripheral vestibular loss
4. Other neurological diagnoses (e.g., peripheral neuropathy, stroke, Parkinson's, central brain lesion)
5. Dizziness due to postural hypotension,
6. Using vestibulosuppressants, antihistamines or ototoxic medications within the previous 3 months will not be included in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Gait Speed- Without Head Turns | 8 week
  The gait speed will be measured using a 10-meter walking test (10MWT). A conventional 10-meter walk course with acceleration and deceleration zones at each end was used to test self-selected walking speed. Individuals in the 10 MWT walk (at a preferred pace) for 10 meters without assistance, with the intermediate 6 meters being timed to allow for acceleration and deceleration. The timing is started when the patient first crosses the 2-meter mark and the timing is stoped when the patient completely passes the 8-meter mark, which allows for 2 meters of acceleration at the start and 2 meters of deceleration at the end of the course. This test will be applied without head turning. A total of 3 trial will be made and the average is recorded in meters per second (m/s).
Gait Speed- With Horizontal Head Turns | 8 week
  The gait speed with horizontal head turns will be measured using a 10-meter walking test (10MWT). A conventional 10-meter walk course with acceleration and deceleration zones at each end was used to test self-selected walking speed. Individuals in the 10 MWT walk (at a preferred pace) for 10 meters without assistance, with the intermediate 6 meters being timed to allow for acceleration and deceleration. The timing is started when the patient first crosses the 2-meter mark and the timing is stoped when the patient completely passes the 8-meter mark, which allows for 2 meters of acceleration at the start and 2 meters of deceleration at the end of the course. The participant will be requested to walk in a pre-measured 10 meter area while performing head turns at approximately 30 degrees towards right and left. A total of 3 trial will be made and the average is recorded in meters per second (m/s).
Gait Speed- With Vertical Head Turns | 8 week
  The gait speed with vertical head turns will be measured using a 10-meter walking test (10MWT). A conventional 10-meter walk course with acceleration and deceleration zones at each end was used to test self-selected walking speed. Individuals in the 10 MWT walk (at a preferred pace) for 10 meters without assistance, with the intermediate 6 meters being timed to allow for acceleration and deceleration. The timing is started when the patient first crosses the 2-meter mark and the timing is stoped when the patient completely passes the 8-meter mark, which allows for 2 meters of acceleration at the start and 2 meters of deceleration at the end of the course. The participant will be requested to walk in a pre-measured 10 meter area while performing head turns at approximately 45 degrees towards up and down. A total of 3 trial will be made and the average is recorded in meters per second (m/s).

SECONDARY OUTCOMES:
Dix Hallpike (Posterior Semicircular Canal Test) | 8 weeks
  The roll test can determine whether the posterior semicircular canal is involved. The patient begins in long-sitting position. Frenzel glasses will be used to visualize the nistagmus during the procedure. The patient will be instructed to rotate his/her head 45 degrees toward the direction of the involed side. With the assistance of the clinician the patient will be quickly bring to lying position with their neck is extended about 45 degrees. Frenzel glasses will be used to visualize the nistagmus for aproximately 60 seconds during the procedure.
Roll Test (Lateral Semicircular Canal Test) | 8 weeks
  The roll test can determine whether the lateral semicircular canal is involved. The roll test requires the person to be in a supine position with their head in 30 degrees of neck flexion. Then the clinician will quickly rotate the head 90 degrees to the left side, and checks for vertigo and nystagmus. Frenzel glasses will be used to visualize the nistagmus for aproximately 60 seconds during the procedure.
Choice Stepping Reaction Time Test | 8 week
  A custom-made Choice Stepping Reaction Time step pad (CSRT-MAT) and a computer unit will be used to evaluate the processing speed. The system is consisted of a CSRT-MAT having pressure-sensitive panels and a display monitor connected to a computer unit. The computer unit recorded the timing of foot lifting and landing. The step direction is indicated by one arrow changing its color. The CSRT device included 2 tests: Stepping Reaction Time (SRT) and Stroop Test (ST). The SRT test will be used in this study. In the SRT test, the participants will be asked to step as quickly as possible onto the corresponding arrow on the CSRT-MAT and then return to the center. The reaction time (RT) measured from stimulus occurrence to movement initiation (lift off), movement time (MT) measured from movement initiation to step finalization (step down) and total response time (RsT) measured as the sum of RT and MT will be recorded.
Fullerton Advanced Balance Scale | 8 week
  The Fullerton Advanced Balance (FAB) scale will be used to evaluate the balance performance of the participants. This performance-based scale consists of 10 test items assessing functional balance (static and dynamic) status. The individual test items are feet together, eyes closed (1), reach forward to retrieve an object (2), turn in a full circle (3), step up and over a bench (4), tandem walk (5), stand on one leg (6), stand on foam, eyes closed (7), two-footed jump (8), walk with head turns (9) and reactive postural control (10). Each test item is scored using a 0-4 scale. The highest score is 40 points, and the lowest is zero. Higher scores indicate better balance abilities.
Nintendo Wii Balance Board- Weight distribution | 8 weeks
  The Nintendo Wii Balance board uses Bluetooth technology and has four pressure sensors that monitor the user's weight and center of balance (the point where an imaginary line drawn vertically through the center of pressure intersects the surface of the Balance Board). This device consists of 4 sensors and a force platform on which these components are placed. Weight distribution will be measured with eyes open and eyes closed on the platform. The right- left and anterior - posterior distribution of weight will be recorded as a percentage.
Dynamic Gait Index | 8 week
  The Dynamic Gait Index (DGI) will be used to assess postural control when walking. The scale assess person's ability to perform various gait tasks such as walking at various speeds, walking with horizontal and vertical head motions, turning while walking, walking over obstacles, turning around obstacles, and stair climbing. The scale consists of eight items, each of which is rated on a scale of 0 to 3. (0 means severe impairment, 3 means normal ability). The optimal DGI score is 24, and subjects with scores of 19 or lower are more likely to fall.
Dizziness Handicap Inventory | 8 week
  The DHI is a 25-item self assessment scale designed to evaluate the self-perceived handicap caused by dizziness. Answers are graded 4 for the response yes, 2 for sometimes, and 0 for no. The scale identifies 3 types of difficulty associated with dizziness: functional difficulties (9 items, representing 36 points in total), emotional difficulties (9 items, 36 points), and physical difficulties (7 items, 28 points). Thus, the scores on the DHI range from 0 (no handicap) to 100 (significant perceived handicap).The total score can be classified as mild (0-30), moderate (>30-60), and severe (>60-100) handicap.
Vestibular Disorders Activities of Daily Living Scale | 8 week
  This scale evaluates the effect of vertigo and balance disorders on independence in routine activities of daily living. Functional (12 questions), ambulation (9 questions), instrumental (7 questions) measures the level of independence in a total of 28 daily living activities. Functional: Includes items on personal care and close relationships, ambulation: items on walking and wandering and instrumental: household chores and hobby activities. In the rating system, it increases from 1 to 10, from being 'independent' to being 'totally dependent'. If the person does not usually do that skill or does not want to respond, he or she marks the "I don't do the activity" section.The sum of the scores of each subsection gives the total score. Functional skills (12-120 points), ambulation skills (9-90 points), instrumental skills (7-70 points) are scored between 28-280 points in total. A low total score indicates the independence of the individual in activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Aytül Özdil, PT, Principal Investigator — Eastern Mediterranean University; Gözde İyigün, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Eyalet/Yerleşke, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iyigun G, Kirmizigil B, Angin E, Oksuz S, Can F, Eker L, Rose DJ. The reliability and validity of the Turkish version of Fullerton Advanced Balance (FAB-T) scale. Arch Gerontol Geriatr. 2018 Sep-Oct;78:38-44. doi: 10.1016/j.archger.2018.05.022. Epub 2018 Jun 4. PMID 29886283
- [Background] Meldrum D, Herdman S, Vance R, Murray D, Malone K, Duffy D, Glennon A, McConn-Walsh R. Effectiveness of conventional versus virtual reality-based balance exercises in vestibular rehabilitation for unilateral peripheral vestibular loss: results of a randomized controlled trial. Arch Phys Med Rehabil. 2015 Jul;96(7):1319-1328.e1. doi: 10.1016/j.apmr.2015.02.032. Epub 2015 Apr 2. PMID 25842051
- [Background] Nada EH, Ibraheem OA, Hassaan MR. Vestibular Rehabilitation Therapy Outcomes in Patients With Persistent Postural-Perceptual Dizziness. Ann Otol Rhinol Laryngol. 2019 Apr;128(4):323-329. doi: 10.1177/0003489418823017. Epub 2019 Jan 4. PMID 30607985
- [Background] Rosiak O, Krajewski K, Woszczak M, Jozefowicz-Korczynska M. Evaluation of the effectiveness of a Virtual Reality-based exercise program for Unilateral Peripheral Vestibular Deficit. J Vestib Res. 2018;28(5-6):409-415. doi: 10.3233/VES-180647. PMID 30714985
- [Background] Yeh SC, Chen S, Wang PC, Su MC, Chang CH, Tsai PY. Interactive 3-dimensional virtual reality rehabilitation for patients with chronic imbalance and vestibular dysfunction. Technol Health Care. 2014;22(6):915-21. doi: 10.3233/THC-140855. PMID 25159998
- [Background] Micarelli A, Viziano A, Augimeri I, Micarelli D, Alessandrini M. Three-dimensional head-mounted gaming task procedure maximizes effects of vestibular rehabilitation in unilateral vestibular hypofunction: a randomized controlled pilot trial. Int J Rehabil Res. 2017 Dec;40(4):325-332. doi: 10.1097/MRR.0000000000000244. PMID 28723718
- [Background] Roettl J, Terlutter R. The same video game in 2D, 3D or virtual reality - How does technology impact game evaluation and brand placements? PLoS One. 2018 Jul 20;13(7):e0200724. doi: 10.1371/journal.pone.0200724. eCollection 2018. PMID 30028839
- [Background] Hsu SY, Fang TY, Yeh SC, Su MC, Wang PC, Wang VY. Three-dimensional, virtual reality vestibular rehabilitation for chronic imbalance problem caused by Meniere's disease: a pilot study<sup/> Disabil Rehabil. 2017 Aug;39(16):1601-1606. doi: 10.1080/09638288.2016.1203027. Epub 2016 Jul 15. PMID 27418422
- [Background] Ozaldemir I, Iyigun G, Malkoc M. Comparison of processing speed, balance, mobility and fear of falling between hypertensive and normotensive individuals. Braz J Phys Ther. 2020 Nov-Dec;24(6):503-511. doi: 10.1016/j.bjpt.2019.09.002. Epub 2019 Sep 23. PMID 31570266